CLINICAL TRIAL: NCT00412490
Title: A Prospective Examination of Smoking Status and Body Image in Surgical Patients With Cancer of the Oral Cavity
Brief Title: Smoking Status and Body Image in Oral Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0126; 5R25CA057730-11 (NIH)
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Oral Cavity Cancer
Keywords: Oral Cavity Cancer; Body Image; Smoking; Appearance; Questionnaire; Interview
MeSH Terms: conditions — Mouth Neoplasms; Smoking | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Smoking Behavior Group: Individuals Having Surgery for Oral Cavity Cancer.
  Interventions: Behavioral: Questionnaire; Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaire — Written survey at 1 Month & 6 Months post surgery.
Behavioral: Interview — One-on-One meeting lasting about one hour, at 1 Month & 6 Months post surgery.

SUMMARY:
Primary Objectives:

1. To characterize smoking behaviors and body image in patients with oral cavity cancer prior to and following surgical procedures.
2. To examine the relationship between smoking status and body image in this sample of head and neck cancer patients.
3. To examine the influence of smoking status and body image on quality of life outcomes.

DETAILED DESCRIPTION:
If you agree to take part in this study, researchers will first perform a test to check the level of carbon monoxide (CO) in your blood. To do this test, you will be asked to blow into a cardboard tube attached to a machine. You will then be asked to fill out some questionnaires and complete a one-on-one interview. All of these things combined will take about an hour to complete. You will be asked basic questions such as your age, education level, and smoking history. You will also be asked questions about your mood, quality of life, and how you feel about your appearance.

If you do not have surgery, your participation in this study will end after this visit. If you have surgery, you will be asked to come back for 2 more study visits, 1 month and 6 months after your surgery. During these evaluations, you will be asked once again to blow into the cardboard tube, fill out questionnaires, and a complete a one-on-one interview. Each visit will last about an hour. You will again be asked questions about your smoking behaviors, mood, quality of life, and how you feel about your appearance. Your participation in this study will be finished after the 6-month evaluation.

This is an investigational study. About 75 people will take part in this research study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Able to provide written informed consent to participate
3. Diagnosis of head and neck malignancy involving an oral cavity site without previous treatment
4. Current treatment plan includes surgical intervention
5. English speaking

Exclusion Criteria:

1. Previous treatment for malignancy in the head and neck region
2. Significant preexisting facial disfigurement from a previous trauma or congenital defect
3. Diagnosis of a serious mental illness involving formal thought disorder (e.g., Schizophrenia) documented in medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals, age 18 years or older, diagnosed with head and neck malignancy involving an oral cavity site without previous treatment, and current treatment plan includes surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2005-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary analysis involve multiple linear regression of body image on gender, age and ethnicity while adjusting for disease and treatment related factors. | Baseline, 1 Month and 6 Months Post Surgery
  Preliminary analyses involve two-sample t-tests of difference in body image between male and female, one-way ANOVA to compare body image across ethnicity groups, and calculation of Pearson product moment correlation coefficients between body image and age.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R. Gritz, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org